CLINICAL TRIAL: NCT00160979
Title: A Study of Transrectal Tumour Oxygen Measurements in Patients With Clinically Localized Prostate Cancer
Brief Title: Transrectal Tumour Oxygen - US Army
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency); Princess Margaret Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UHN REB 00-0443-C; US Army DAMD17-01-1-0111
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms

ARMS (1):
- hypoxia and RT in prostate cancer (Experimental)
  Interventions: Procedure: Pre-treatment tumour oxygen measurements

INTERVENTIONS:
Procedure: Pre-treatment tumour oxygen measurements — Pre-treatment tumour oxygen measurements

SUMMARY:
Prostate cancer is now the most commonly diagnosed tumor among men in the United States. Most patients have tumors that are confined to the prostate gland at diagnosis and are suitable for treatment with surgery or radiotherapy (RT) that is aimed at curing the disease. Nevertheless, despite recent improvements in these treatments, a large number of men continue to die of prostate cancer. These patients often have spread of tumor to other areas of the body, and are treated with hormones that produce initial tumor shrinkage. However, over time the tumor learns to grow despite continued hormonal treatment. Effective therapy for patients with hormone-resistant prostate cancer is lacking and patients often deteriorate quickly and die. Thus, there is a need for better treatment that cures prostate cancer at an early stage, and a better understanding of the biology of prostate cancer specifically with respect to factors that determine the effectiveness of RT, the spread of tumor and the development of hormone-resistant disease.

Low levels of oxygen (hypoxia) are known to exist in many human tumors, and studies have shown that hypoxic tumors are less likely to be cured by RT. In addition, hypoxia may lead to lower cure rates following surgery, spread of cancer to other areas of the body, and changes in the genetic characteristics of the cancer cells that cause them to behave more aggressively.

The importance of hypoxia in prostate cancer has not previously been evaluated. The aims of this study are to determine how often hypoxia occurs in early prostate cancer and whether hypoxia influences the success of RT, tumor spread beyond the prostate to bones and other organs and the development of hormone-resistant disease. Patients will have tumor oxygen levels measured using a special fine-needle electrode system prior to beginning treatment with either RT or the combination of hormones plus RT. The measurements will be made through the rectum using ultrasound to position and guide the electrode. A biopsy of the tumor will be obtained at the site of the measurements, and this will be used to determine how oxygen influences changes in the genetic character of prostate cancer cells. A total of 195 patients will be evaluated in this way over 3 years.

This study will provide unique information about the behavior of prostate cancer, which may help explain why currently available treatments including surgery, RT and hormones fail to cure patients. Assuming that this study shows hypoxia to be important in prostate cancer, future work will focus on new anti-hypoxia treatments to be used in combination with surgery or RT with the aim of overcoming this obstacle and improving cure rates.

ELIGIBILITY:
Inclusion Criteria:

* A histologic diagnosis of adenocarcinoma of the prostate
* A decision to treat using high-dose conformal radiotherapy, with or without neoadjuvant and concurrent androgen ablation
* Clinical stage T2a or T2b, N0, M0 (UICC 1997 68)
* No hormonal or cytotoxic anti-cancer therapy prior to study entry
* ECOG performance status of 2 or less
* Ability to understand the English language
* Signed informed consent

Exclusion Criteria:

* Patients with prior or active malignancy within 5 years of the diagnosis of prostate cancer, except non-melanoma skin cancer

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Estimated)
Dates: Start 2001-01; Primary Completion 2023-02 (Actual); Study Completion 2023-02 (Actual)

PRIMARY OUTCOMES:
To determine the relationship between pre-treatment prostate cancer oxygen levels and long-term disease control following treatment with radiotherapy, and the independent prognostic effect of oxygen measurements. | after follow-up is completed
To determine the relationship between pre-treatment tumor oxygen levels and mutations of the p53 gene, and the impact of this interaction on patient outcome. | after follow up is completed

SECONDARY OUTCOMES:
To evaluate oxygen levels in clinically localized prostate cancer prior to treatment. | after follow-up is completed
To determine the relationship between pre-treatment tumor oxygen levels and the subsequent development of metastases and androgen-resistant prostate cancer. | after follow is completed
To determine whether androgen ablation overcomes any adverse effect of hypoxia on outcome. | after follow up is completed

CONTACTS AND LOCATIONS:
Overall Officials: Michael Milosevic, MD, Principal Investigator — Princess Margaret Hospital, Canada
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada